CLINICAL TRIAL: NCT04197791
Title: Effect of Core Stabilization Exercises and Neuromuscular Electrical Stimulation (NMES) in Patients With Idiopathic Pulmonary Fibrosis (IPF) Randomized Controlled Trial
Brief Title: Effect of Core Stabilization Exercises and Neuromuscular Electrical Stimulation in Patients With Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, ELÇİN ÇAKIR, MSc student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 272303
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Core Stabilization Exercises
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation (NMES) (Experimental): Neuromuscular Electrical Stimulation will be applied to 18 patients with idiopathic pulmonary fibrosis. The application time will be 30 minutes. Treatment will be programmed for 2 days per week. The program will continue for 6 weeks.
  Interventions: Device: Neuromuscular Electrical Stimulation
- Core Stabilization Exercises (Experimental): Core stabilization exercises will be applied to 18 patients with idiopathic pulmonary fibrosis. The exercise time will be 30 minutes. Treatment will be programmed for 2 days per week. The program will continue for 6 weeks.
  Interventions: Other: Core Stabilization Exercises

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation(NMES) to core stabilization muscles will be applied using 8 electrodes. The application time will be 30 minutes. Treatment will be programmed for 2 days per week. The program will continue for 6 weeks.
  Arms: Neuromuscular Electrical Stimulation (NMES)
Other: Core Stabilization Exercises — Warm-up and cool-down exercises will be performed before and after core stabilization exercises. The exercise time will be 30 minutes. Treatment will be programmed for 2 days per week. The program will continue for 6 weeks.
  Arms: Core Stabilization Exercises

SUMMARY:
Interstitial lung disease (ILD) refers to various diseases that occur idiopathic or secondary to some causes, commonly affecting the lung parenchyma, and present with varying degrees of inflammation and fibrosis. Idiopathic pulmonary fibrosis (IPF) progressing with progressive shortness of breath causes a decrease in exercise capacity and quality of life, restrictive changes in pulmonary function tests and a decrease in diffusion capacity. It has been reported that core stabilization exercises improve respiratory function, respiratory muscle strength and functional capacity in healthy individuals and some disease groups. It has also been reported that neuromuscular electrical stimulation (NMES) applied to lower extremity, upper extremity and back or quadriceps muscles reduces dynamic hyperinflation and dyspnea during exercise and increases exercise capacity in COPD patients.No studies have been performed using core stabilization exercises and NMES in IPF patients. It can be assumed that this therapeutic intervention may also be useful in IPF.

Our study was planned to investigate the efficacy of core stabilization exercises and NMES in patients with IPF.

DETAILED DESCRIPTION:
Stable idiopathic pulmonary fibrosis will be included in the study from the Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital. Patients will be randomized into 2 groups; Neuromuscular Electrical Stimulation (NMES) and Core Stabilization Exercises Training Group (n: 18): 2 days per week for 6 weeks duration. The demographic measurements, respiratory function test, respiratory muscle strength, dyspnea, 6 minutes walking test, quality of life, depression and clinical characteristics and physical fitness of the patients will be recorded. The following parameters will be evaluated before and after the training of the patients in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Having no infection or exacerbation in the last 3 months
* Having no uncontrolled cardiological, psychological problems
* Having no neoplasm, sarcoidosis or collagen vascular diseases
* Having no neurological, inner ear or orthopedic disease
* Patients who volunteered to study

Exclusion Criteria:

* Over 75 years,
* Chronic obstructive pulmonary disease (COPD)
* Acute coronary artery disease,
* Collagen vascular disease,
* Pneumoconiosis,
* Sarcoidosis,
* Cancer
* Non-parenchymal restrictive lung disease and other serious comorbid conditions,
* Oxygen saturation in room air at rest <80%
* During acute exacerbation,
* Echocardiography RVSP> 50 mmHg
* Patients taking more than 20mg corticosteroid per day
* Contraindications to apply the neuromuscular electrical stimulation (pace maker, sensory defects, etc...)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline and 6 weeks
  Change from baseline Forced Vital Capacity (FVC) in respiratory function test at 6 weeks. FVC will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Forced Expiratory Volume 1 second (FEV1) | Baseline and 6 weeks
  Change from baseline Forced Expiratory Volume 1 second (FEV1) in respiratory function . FEV1 will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Forced Expiratory Volume 1 second / Forced Vital Capacity (FEV1 / FVC) | Baseline and 6 weeks
  Change from baseline FEV1 / FVC in respiratory function test at 6 weeks. FEV1 / FVC will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Forced Expiratory flow from between 25% to 75% of Vital Capacity (FEF 25-75) | Baseline and 6 weeks
  Forced expiratory flow at 25-75% of FVC [FEF25-75] (L/sec) was measured with lung spirometry as it was described for FVC, FEV1, FEV1 / FVC measurements.
Peak flow rate (PEF) | Baseline and 6 weeks
  Change from baseline Peak flow rate (PEF) in respiratory function test at 6 weeks. PEF will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Single-breath Diffusing Capacity for Carbon Monoxide (DLCO) | Baseline and 6 weeks
  The DLCO is a pulmonary function test that measures the capacity for the lung to carry out gas exchange between the inhaled breath and the pulmonary capillary blood vessels and the DLCO %-predicted represents the DLCO expressed as a percentage of the expected normal valued based on the participant's age, height, gender and ethnicity. The DLCO %-predicted is reduced in patients with interstitial lung disease and is used as a measure of disease severity.
Functional capacity | Baseline and 6 weeks
  Change from baseline functional capacity test at 6 weeks. Functional capacity will be assessed by the 6 minute walking test. The test will be performed according to American Thoracic Society (ATS) criteria. Patients will be allowed to rest for 10 minutes before the test. Heart rate, blood pressure, respiratory frequency, oxygen saturation, fatigue and dyspnea perception will be recorded before and after the test. Walking distance will be calculated.

SECONDARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) | Baseline and 6 weeks
  Change from baseline Maximum Inspiratory Pressure (MIP) at 6 weeks. Respiratory muscle strength will be measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The most commonly used method for evaluating respiratory muscles is MIP measurement is a non-invasive technique.
Maximum Expiratory Pressure (MEP) | Baseline and 6 weeks
  Change from baseline Maximum Expiratory Pressure (MEP) at 6 weeks. Respiratory muscle strength will be measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The most commonly used method for evaluating respiratory muscles is MEP measurement is a non-invasive technique.
Physical Activity | Baseline and 6 weeks
  Change from baseline physical activity scores at 6 weeks. International Physical Activity Questionnaire (IPAQ) - Short Form (Turkish version of scale ).This questionnaire assesses, in minutes, the physical activity performed by the volunteers during the period of one week. The IPAQ considered all activities carried out by the volunteer (e.g. leisure, sport, exercise, and activities at home or in the garden). According to the responses, the volunteer is considered very active, active, irregularly active or sedentary, according to the intensity and time of the exercises practiced over the last week.
Change from baseline quality of life: King's Brief Interstitial Lung Disease Questionnaire (K-BILD) | Baseline and 6 weeks
  Quality of life will be measured with King's Brief Interstitial Lung Disease Questionnaire (K-BILD). It is a 15-item validated questionnaire assessing health status in patients with an interstitial lung disease. Questions are related to three domains: breathlessness and activities, psychological aspects, and chest symptoms. Each question has 7 possible answers. The questionnaire has a scale from 0 - 100, in which 100 means highest quality of life.
Change from baseline quality of life: Hospital Anxiety and Depression Scale (HADS) | Baseline and 6 weeks
  Quality of life will be measured with the Hospital Anxiety and Depression Scale (HADS). It is a 14-item questionnaire, 7 items are related to depression and 7 items are related to anxiety. Each question has 4 different answer options, each scored from 0-3. Scores are summed up for each field (depression or anxiety) with 0 points as lowest possibility and 21 scores as highest (0-7 = normal, 8-10 = borderline abnormal, and 11-21 = abnormal).
The Fatigue Severity Scale | Baseline and 6 weeks
  The Fatigue Severity Scale is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Respondents answer using a Likert scale ranging from 1 to 7. ''1'' indicates strong disagreement with the statement, while ''7'' indicates strong agreement. Total score is calculated by deriving an arithmetic mean. FSS scores range from 0-63. A score of 36 or higher generally indicates severe fatigue.
Timed up and go test | Baseline and 6 weeks
  Functional mobility was measured with Timed up and go test [TUGT] (sec). The patient sitting on chair stood up with the instruction of physiotherapist and walked 3 meters as fast as possible, walked back to the chair and sat down again. The total duration was recorded in seconds. Lower time reflects better functional mobility. TUGT was performed with 3 repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Vainshelboim B, Oliveira J, Yehoshua L, Weiss I, Fox BD, Fruchter O, Kramer MR. Exercise training-based pulmonary rehabilitation program is clinically beneficial for idiopathic pulmonary fibrosis. Respiration. 2014;88(5):378-88. doi: 10.1159/000367899. Epub 2014 Oct 23. PMID 25341682
- [Background] Park M, Seok H, Kim SH, Noh K, Lee SY. Comparison Between Neuromuscular Electrical Stimulation to Abdominal and Back Muscles on Postural Balance in Post-stroke Hemiplegic Patients. Ann Rehabil Med. 2018 Oct;42(5):652-659. doi: 10.5535/arm.2018.42.5.652. Epub 2018 Oct 31. PMID 30404414
- [Background] Mustafaoglu R, Demir R, Demirci AC, Yigit Z. Effects of core stabilization exercises on pulmonary function, respiratory muscle strength, and functional capacity in adolescents with substance use disorder: Randomized controlled trial. Pediatr Pulmonol. 2019 Jul;54(7):1002-1011. doi: 10.1002/ppul.24330. Epub 2019 Apr 26. PMID 31026384